CLINICAL TRIAL: NCT05975892
Title: Transplantation of Bone Marrow Mesenchymal Stromal Cells for Bone Regeneration in Periodontal Disease
Brief Title: Transplantation of Bone Marrow Mesenchymal Stromal Cells for Periodontal Regeneration
Acronym: BMMSC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto Venezolano de Investigaciones Cientificas (Other)
Collaborators: Universidad Central de Venezuela (Other); Hospital Central Dr. Plácido D. Rodriguez Rivero, San Felipe, Yaracuy (Unknown)
Responsible Party: Principal Investigator, Dylana Diaz Solano, Clinical Investigator, Instituto Venezolano de Investigaciones Cientificas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IVIC-UTC-MSC-Periodontal
Record Dates: First submitted 2023-07-14; First posted 2023-08-04 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-07

CONDITIONS: Chronic Periodontal Disease; Aggressive Periodontitis
Keywords: Mesenchymal stromal cells; Periodontal regeneration; Bone regeneration; Periodontitis
MeSH Terms: conditions — Chronic Periodontitis; Aggressive Periodontitis; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic MSCs transplantation in periodontal disease (Experimental): Allogeneic MSC harvested and cultured in osteogenic medium are seeded on collagen scaffold, mixed with autologous platelet rich plasma clot. The MSCs construct (MSCs/Coll/PRP clot) is implanted in the bone defect.
  Interventions: Biological: Transplantation of allogeneic MSCs in periodontal disease

INTERVENTIONS:
Biological: Transplantation of allogeneic MSCs in periodontal disease — Oral surgery is performed in patients with periodontal disease, under local anesthesia. An incision will be made on the periodontal lesion, A full-thickness flap is elevated on both the buccal and lingual areas and the inner epithelium of the flap removed. Granulation tissue is removed from bone defect area, and a root planning is performed. MSC construct is placed around the bone defect and a collagen membrane is used to cover and close off the bone defect site. The flap will be repositioned and the wound closed by a suture

SUMMARY:
The goal of this study is to evaluate the capacity of allogeneic bone marrow mesenchymal stromal cells (MSC) to induce bone regeneration in patients with periodontal disease. MSC cultured are loaded on a collagen scaffold, included into autologous platelet rich plasma clot and implanted in the bone defect.

DETAILED DESCRIPTION:
The clinical protocol is designed to evaluate the bone regeneration capacity of allogeneic MSCs for the treatment of patients with chronic or aggressive periodontal disease. Patients with either a 2- or 3-wall intrabony defects are included in this study. A bioengineering construct, constituted by allogeneic MSCs and a collagen scaffold, is incorporated into platelet rich plasma (PRP) clot, which is implanted at the bone defect site. Follow up of treated tooth are assessed by clinical evaluation, intraoral radiography and cone-beam CT.

ELIGIBILITY:
Inclusion Criteria:

* Medical healthy
* Minimum age of 18 years old
* Diagnosis of chronic or aggressive periodontitis
* Vertical intrabony defects of three or two walls
* PPD >= 5 mm
* Radiographic evidence of alveolar bone loss of at least 3 mm
* Minimim 20 teeth presents in mouth.
* Informed consent of the patient

Exclusion Criteria:

* Smoking
* Pregnancy or lactating
* Receiving immunosuppressive drugs, anticoagulants, antibiotics or analgesic drugs
* Diabetics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-08-30 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in clinical attachment level (CAL) | Follow-up includes evaluation at 3, 6, 9 and 12 months post-transplantation
  Expressed as the distance in millimeters from the cemento-enamel junction (CEJ) to the bottom of the probable gingival/periodontal pocket.
Change in probing pocket depth (PPD) | Follow-up includes evaluation at 3, 6, 9 and 12 months post-transplantation
  The distance from the gingival margin to the bottom of the gingival sulcus/pocket, is measured by means of periodontal probe.
Gingival recession (GR) | Follow-up includes evaluation at 3, 6, 9 and 12 months post-transplantation
  Exposure of the tooth through apical migration of the gingiva will be recorded as the distance in millimeters from the CEJ to the gingival margin
Change in bone density | Follow-up includes evaluation at 3, 6, 9 and 12 months post-transplantation
  Changes in the density of the periodontal bone defect will be detected by Cone beam Tomography
Change in Tooth Mobility (TM) | Follow-up includes evaluation at 3, 6, 9 and 12 months post-transplantation
  Changes from baseline in tooth mobility will be recorded.
Change in bone depth | Follow-up includes evaluation at 3, 6, 9 and 12 months post-transplantation
  The vertical bone defects will be assessed by X-rays. The postoperative depth of the intrabony defect will be calculated from the distance between the cemento-enamel junction and the bone crest on the preoperative and postoperative radiographs at the same magnification.

CONTACTS AND LOCATIONS:
Overall Officials: Jose E Cardier Montalvo, MD, PhD, Principal Investigator — Instituto Venezolano de Investigaciones Cientificas
Locations (1):
- Instituto Venezolano de Investigaciones Cientificas, Caracas, Miranda, Venezuela

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wittig O, Diaz-Solano D, Cardier J. Viability and functionality of mesenchymal stromal cells loaded on collagen microspheres and incorporated into plasma clots for orthopaedic application: Effect of storage conditions. Injury. 2018 Jun;49(6):1052-1057. doi: 10.1016/j.injury.2018.04.005. Epub 2018 Apr 5. PMID 29678307
- [Background] Wittig O, Romano E, Gonzalez C, Diaz-Solano D, Marquez ME, Tovar P, Aoun R, Cardier JE. A method of treatment for nonunion after fractures using mesenchymal stromal cells loaded on collagen microspheres and incorporated into platelet-rich plasma clots. Int Orthop. 2016 May;40(5):1033-8. doi: 10.1007/s00264-016-3130-6. Epub 2016 Mar 16. PMID 26980620
- [Background] Gomez M, Wittig O, Diaz-Solano D, Cardier JE. Mesenchymal Stromal Cell Transplantation Induces Regeneration of Large and Full-Thickness Cartilage Defect of the Temporomandibular Joint. Cartilage. 2021 Dec;13(1_suppl):1814S-1821S. doi: 10.1177/1947603520926711. Epub 2020 Jun 4. PMID 32493042
- [Background] Gomez-Sosa JF, Diaz-Solano D, Wittig O, Cardier JE. Dental Pulp Regeneration Induced by Allogenic Mesenchymal Stromal Cell Transplantation in a Mature Tooth: A Case Report. J Endod. 2022 Jun;48(6):736-740. doi: 10.1016/j.joen.2022.03.002. Epub 2022 Mar 18. PMID 35307516